CLINICAL TRIAL: NCT07101341
Title: Analysis of the Acute Effects of Aerobic Exercise and High-intensity Interval Exercise, With and Without the Simultaneous Application of Immersive Virtual Reality
Brief Title: Acute Effects of Aerobic Exercise and High-intensity Interval Exercise With Immersive Virtual Reality
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Adrián Escriche Escuder, Assistant professor, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-FIS-3483189
Record Dates: First submitted 2025-07-22; First posted 2025-08-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Acute Effects of Exercise in Healthy People; Health Adult Subjects
Keywords: virtual reality; immersive virtual reality; exergame
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Traditional aerobic exercise (Experimental)
  Interventions: Procedure: Traditional aerobic training
- High-intensity interval training (Experimental): A single session of exercise
  Interventions: Procedure: High Intensity Interval Training (HIIT)
- Aerobic exercise applied with reality virtual (Experimental): A single session of exercise
  Interventions: Procedure: Aerobic training performed with a immersive virtual reality application
- High-intensity interval training applied with virtual reality (Experimental): A single session of exercise
  Interventions: Procedure: High Intensity Interval Training (HIIT) performed with a immersive virtual reality application

INTERVENTIONS:
Procedure: Traditional aerobic training — 5 minutes of warm-up at increasing intensity up to 60% of maximum heart rate (HRmax) + 20 minutes between 60-80% of HRmax + 5 minutes of cool-down at decreasing intensity (30-60% HRmax)
  Arms: Traditional aerobic exercise
Procedure: High Intensity Interval Training (HIIT) — 5 minutes warm-up at increasing intensity up to 60% maximum heart rate (HRmax) + 20 minutes main part consisting of 10 repetitions of the combination of 1 minute at 75-90% HRmax and 2 minutes of active rest with light pedaling (50% HRmax) + 5 minutes cool-down at decreasing intensity (30-60% HRmax)
  Arms: High-intensity interval training
Procedure: Aerobic training performed with a immersive virtual reality application — 5 minutes of warm-up at increasing intensity up to 60% Maximum heart rate (HRmax) + 20 minutes between 60-80% of HRmax + 5 minutes of cooling at decreasing intensity (30-60% HRmax), with the use of virtual reality glasses and an immersive virtual reality application
  Arms: Aerobic exercise applied with reality virtual
Procedure: High Intensity Interval Training (HIIT) performed with a immersive virtual reality application — 5 minutes warm-up at increasing intensity up to 60% Maximum heart rate (HRmax) + 20 minutes main part consisting of 10 repetitions of the combination of 1 minute at 75-90% HRmax and 2 minutes of active rest with light pedaling (50% HRmax) + 5 minutes cool-down at decreasing intensity (30-60% HRmax), with the use of virtual reality glasses for an immersive virtual reality application
  Arms: High-intensity interval training applied with virtual reality

SUMMARY:
This study aims to compare the acute effects at the cardiovascular (heart rate, blood pressure) and physiological (lactate) levels, as well as the perception of effort and fatigue, of four exercise modalities, one based on the traditional aerobic training methodology, another based on high-intensity interval training (HIIT), another consisting of aerobic exercise performed in conjunction with an immersive virtual reality (VR) application, and a last one consisting of exercise with HIIT-type parameters but also performed in conjunction with an immersive VR application.

All participants will complete one session of each of the four exercise modalities, analyzing the variables studied in each for subsequent analysis and comparison.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people between 18 and 35 years old

Exclusion Criteria:

* Current or recent injury that affects training
* Condition that prevents exercise (decompensated heart disease, decompensated respiratory disease, significant mobility difficulties, etc.)
* Visual problems that prevent exercise with virtual reality headsets

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Blood lactate | During the 5 minutes after finishing the exercise session of each intervention modality (Days 1, 8, 15 and 22 from the start of the study)
  Analysis of blood lactate concentration

SECONDARY OUTCOMES:
Heart rate pattern | During each exercise session (Days 1, 8, 15 and 22 from the start of the study)
  Heart rate pattern, measured with a heart rate monitor
Systolic and diastolic blood pressure | During the 5 minutes after finishing the exercise session of each intervention modality (Days 1, 8, 15 and 22 from the start of the study)
  Systolic and diastolic blood pressure, measured with a sphygmomanometer
Perception of effort | During the first minute after finishing the exercise session of each intervention modality (Days 1, 8, 15 and 22 from the start of the study)
  Individual perception of effort during exercise, assessed with a modified Borg scale (0-10), where 0 is "no effort" and 10 corresponds to the "maximum possible perception of effort".
Perception of fatigue | During the first minute after finishing the exercise session of each intervention modality (Days 1, 8, 15 and 22 from the start of the study)
  Individual perception of fatigue, with a numerical scale from 0 to 10, where 0 is "no fatigue" and 10 corresponds to the "maximum perception of fatigue possible"
Physical performance | During the 5 minutes after finishing the exercise session of each intervention modality (Days 1, 8, 15 and 22 from the start of the study)
  Physical performance, assessed by calculating the sets, repetitions and kg mobilized during the exercise time.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Escriche-Escuder, PhD, Principal Investigator — University of Valencia
Locations (1):
- Faculty of Physiotherapy, University of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study will be available from the corresponding author upon reasonable request.